CLINICAL TRIAL: NCT01524354
Title: Monitoring of Anesthetic Depth During Surgical Correction of Acquired Valvular Disorders
Brief Title: Depth of Anesthesia in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Depth-28
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Heart Valve Diseases
Keywords: depth of anesthesia; valve surgery
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients received maintenance of anesthesia with continuous infusion of propofol according to recommendations of the manufacturer.
  Interventions: Procedure: maintenance of anesthesia
- cerebral state index (Active Comparator): Patients received continuous infusion of propofol with rate maintaining cerebral state index (CSI) between 40 and 60 points.
  Interventions: Procedure: maintenance of anesthesia

INTERVENTIONS:
Procedure: maintenance of anesthesia — intraoperative maintenance of anesthesia with propofol under control of cerebral state index at 40-60 points
  Other Names: Controlled anesthesia depth
  Arms: cerebral state index
Procedure: maintenance of anesthesia — intraoperative maintenance of anesthesia with propofol according to recommendations of the manufacturer
  Other Names: Controlled anesthesia depth
  Arms: Control

SUMMARY:
The aim of our study was to evaluate the significance of monitoring anesthetic depth for the conduct of anesthesia and the early postoperative period in patients subjected to surgical correction of combined valvular disorders.

DETAILED DESCRIPTION:
Our aim was to evaluate the effect of monitoring anesthetic depth on duration of postoperative mechanical ventilation and ICU stay after surgical correction of combined valvular disorders.

ELIGIBILITY:
Inclusion Criteria:

* requirement of surgical correction of two or more valves

Exclusion Criteria:

* no

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
duration of postoperative mechanical ventilation | 24 hours postoperatively
  Criteria for termination of postoperative respiratory support were the following: patient able to cooperate; adequate muscular tone; SpO2 > 95% with FiO2 0.5; PaCO2 < 45 mm Hg; postoperative bleeding rate < 50 mL hr-1; stable hemodynamics without inotropic/vasopressor support; body temperature of > 35 °C. Temporary pacing was not regarded as a contraindication for tracheal extubation.

SECONDARY OUTCOMES:
length of ICU stay | 7 days postoperatively
  The time until 'fit for ICU discharge' criteria as well as the actual length of the ICU stay were registered. The 'fit for ICU discharge' criteria included the following: fully oriented patient, SaO2 > 90% on room air, no episodes of severe arrhythmias, bleeding < 50 mL hr-1, diuresis > 0.5 mL kg-1 hr-1, no need for inotropic/vasopressor support and no signs of ischemia on ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, MD, PhD, Study Director — Northern State Medical Univercity